CLINICAL TRIAL: NCT00505947
Title: Infliximab for Diabetic Macular Edema Refractory to Laser Photocoagulation: a Randomized, Double-Masked, Placebo-Controlled, Cross-Over, 32 Weeks Study
Brief Title: Treatment of Refractory Diabetic Macular Edema With Infliximab
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The number of the anticipated participants was not achieved
Sponsor: University of Athens (Other)
Responsible Party: Petros Sfikakis, University of Athens
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C0168X97; EU-0129
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Diabetic Macular Edema; Visual Acuity; Diabetic Retinopathy
Keywords: macular edema; diabetes mellitus; visual loss; diabetic retinopathy; macula; maculopathy; infliximab
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Diabetes Mellitus; Vision Disorders; Macular Degeneration | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Infliximab 5 mg/Kg body weight by intravenous infusion on visit 1 (week 0), visit 2 (week 2), visit 3 (week 6)and visit 5 (week 14).
  Afterwards, after a washout period of 2 weeks, arm A will receive placebo at visits 6 (week 16), visit 7 (week 18), visit 8 (week 22)and visit 30 (week 30)
  Interventions: Drug: infliximab; Drug: placebo
- B (Placebo Comparator): Arm B will receive placebo at visit 1 (week 0), visit 2 (week 2), visit 3 (week 6)and visit 5 (week 14).
  Afterwards, after a washout period of 2 weeks, group B will receive infliximab 5 mg/Kg body weight by intravenous infusion at visit 6 (week 16), visit 7 (week 18), visit 8 (week 22)and visit 30 (week 30)
  Interventions: Drug: infliximab; Drug: placebo

INTERVENTIONS:
Drug: infliximab — infliximab 5 mg/Kg body weight by intravenous infusion
  Other Names: Remicade
Drug: placebo — placebo 5 mg/Kg body weight by intravenous infusion
  Other Names: placebo: a solution of similar appearance with infliximab

SUMMARY:
The purpose of this study is to determine if treatment with infliximab improves macular edema which is refractory to laser photocoagulation in patients with diabetes.

DETAILED DESCRIPTION:
Retinopathy affects on average 30% of all patients with diabetes. Good glycaemic control delays the onset and progression of retinopathy in subjects with both type 1 and type 2 diabetes. However, the incidence of retinopathy has not been declining in type 1 diabetes over the last decades, even if visual acuity may be better preserved. As many as 20% of the patients with type 2 diabetes mellitus have already retinopathy at the time of diagnosis of diabetes. Diabetic macular edema (DME) is a serious manifestation of diabetic retinopathy that produces loss of central vision. Data from the Wisconsin Epidemiological Study of Diabetic Retinopathy (WESDR) estimate that after 15 years of known duration of diabetes the prevalence of DME is 20% in patients with type 1 diabetes mellitus, 25% in patients with type 2 diabetes who are treated with insulin, and 14% in the patients with type 2 diabetes who are not treated with insulin. Concerning the natural history a previous study has shown that 53% of the eyes with DME involving the centre of the macula, lost two or three lines of visual acuity over a two year period. In addition, in the Early Treatment Diabetic Retinopathy Study (ETDRS), 33% of untreated eyes available for follow-up at the 3-year visit, all with oedema involving the centre of the macula at baseline, had experienced a 15 or more letter decrease in visual acuity score.

The federal budgetary cost of blindness was estimated to be $4.1 billion in the U.S. for the year 1990, and 97% of these costs were accounted for by the working-age adult group. Health care and economic burdens are further compounded by the resulting decline in quality of life; thus, the true impact on society cannot be estimated on a monetary basis alone.

Although the etiology of DME is unclear, an altered local expression of the pleiotropic cytokine tumor necrosis factor (TNF) may play an important role in pathogenesis. Standard treatment of clinically significant DME (i.e. reduction of visual acuity due to DME) consists of laser photocoagulation (two sessions for optimal results?). However, this treatment effectively reduces the risk of vision loss in only 50% of cases. Even among those patients who achieve an initial response recurrences are common, requiring ongoing treatment. Vitreomacular traction or the vitreous itself may play a role in increased retinal vascular permeability. Removal of the vitreous or relief of mechanical traction with pars plana vitrectomy and membrane stripping may be followed by substantial resolution of macular edema and improvement in visual acuity. However, this treatment may be applicable only in specific subset of eyes with DME. It also requires a complex surgical intervention with its inherent risks, recovery time and expenses. Other treatment modalities such as pharmacologic therapy with oral protein kinase C inhibitors, antibodies targeted at vascular endothelial growth factor (VEGF), intravitreal corticosteroid injection, or high doses of non-steroidal anti-inflammatory agents that lower retinal expression of TNF are under investigation.

Infliximab is a chimeric IgG1 monoclonal antibody with an approximate molecular weight of 149,100 Dalton. It is composed of human constant and murine variable regions. Infliximab binds specifically to human tumour necrosis factor alpha (TNF-a) with an association constant of 1010 M-1. Infliximab is produced by a recombinant cell line cultured by continuous perfusion and is purified by a series of steps that includes measures to inactivate and remove viruses.

Infliximab is currently used for the treatment of inflammatory arthritic conditions and inflammatory disease with a favorable safety profile. Because of the limitations of current treatments for DME, and based on our recent findings indicating that infliximab is an effective therapy for cystoid ME associated with uveitis, we decided to assess whether infliximab is effective for patients with diabetes (type 1 or 2) and sight-threatening DME.

We have found that a clinically meaningful anatomic and functional improvement was achieved after two infliximab infusions in 4 of 6 eyes with severe diffuse DME (i.e. macular thickness >400 μm); in contrast the remaining 2 eyes with coexisting epiretinal membranes did not improve. The observed recovery of useful vision represents a very significant clinical result, especially for those eyes in which DME was refractory to laser photocoagulation. Comparable beneficial results have been obtained in our patients with severe, chronic cystoid ME complicating intermediate uveitis, Adamantiades-Behcet's disease, or adult type vascular pseudotumor. Repeated treatment in one diabetic patient produced a further significant improvement of DME, indicating that the clinical response to anti-TNF dosing regimens is individualized, as it has also been observed in patients with arthritis, or in patients with uveitic ME. Thus, a sustained beneficial effect of infliximab for DME may require long-term treatment. Infliximab was well tolerated by our patients in all studies conducted at our site.

Results from a preliminary study suggest a central role for TNF-mediated pathogenesis mechanisms in DME. Recent experimental evidence also indicates that low-grade subclinical inflammation is responsible for many of the signature vascular lesions of diabetic retinopathy On the other hand, studies in patients with arthritis have shown that anti-TNF therapy negatively affects vascular permeability and angiogenesis by decreasing the potent angiogenic vascular endothelial growth factor, which has been implicated directly in the pathogenesis of DME and diabetic retinopathy.

Four women, aged 52 to 76 years, with type 2 diabetes who were in danger of vision loss due to severe DME were included in this prospective, non-comparative case series. They all used oral antidiabetic agents for 14 to 20 years, while one patient required exogenous insulin therapy for the last 4 years. Patients were free of other major medical disorders and they had no evidence of infection. Following full discussion and after obtaining informed consent, 2 infusions of infliximab (5mg/kg, Remicade, Schering-Plough, Greece) with one month interval, were given intravenously over 3 hours in an outpatient setting on a compassionate basis. Additional infusions were offered in 3 patients. Concomitant medications remained unchanged.

Complete ophthalmic examination and Optical Coherence Tomography (OCT, Model 3000, Zeiss, Humphrey Systems) were performed immediately before each infliximab infusion, as well as 2 months after the last infusion. The main outcome measurements were best corrected visual acuity (BCVA) and macular thickness. The OCT-derived maximum height of DME was recorded as described previously in detail. The student t-test for paired data was used to compare logarithm of minimum angle of resolution (logMAR) transformed BCVA, as well as macular thickness between baseline and post-treatment.

DME was present in 7 eyes, 6 of which were refractory to previous treatment with laser photocoagulation. DME was classified as severe in 6 eyes (range of macular thickness 420-720 μm) and as mild in 1 eye (macular thickness of 290 μm after vitrectomy). A dense epiretinal membrane was present in 2 eyes with severe DME. BCVA at baseline was profoundly impaired, ranging from 'hand motion' to 0.1 at the Snellen chart. At one month after the first infliximab infusion, macular thickness had decreased in 5 from 7 eyes from [mean(SD)]503 (171) to 426 (165) μm (p=0.033). The 2 eyes with coexisting epiretinal membranes did not improve. Two months after the second infusion, the macular thickness had further regressed to 330 (134) μm (range 170 to 515 μm, p=0.028, compared to baseline). The BCVA was increased in all 5 eyes from a baseline mean at the Snellen chart of 0.03 to 0.15 (logMAR 1.42 (0.45) to 0.82 (0.27), p=0.01).

At 3 months post-baseline a third infliximab infusion was offered in those 3 patients who had the least improvement of DME. Repeated OCT after 2 months revealed a further decrease of macular thickness in 3 of 5 eyes, by 7 %, 15 % and 23 %, respectively. At this point the patient who still had the most severe condition received a fourth infliximab infusion; remarkably, a repeated OCT two months later revealed a marked resolution of severe DME, while BCVA had improved from counting fingers at baseline to 0.2. Infliximab therapy was well tolerated and no ocular or extra-ocular side effects were noted. In further available follow-up ranging from 4 to 7 months post-treatment, a recurrence of DME was observed in 2 of 5 eyes, albeit at a less severe level.

For detailed information about the safety of infliximab please refer to summary of product characteristics. Active tuberculosis may develop soon after the initiation of treatment with infliximab. Before prescribing the drug, physicians should screen patients for latent tuberculosis infection or active disease.

Based on the above, we believe that administration of infliximab may be a reasonable therapeutic approach in diabetic patients who are in danger of vision loss due to refractory DME. Therefore, a controlled study on the safety and efficacy of infliximab treatment in DME refractory to laser photocoagulation is warranted. Because of our preliminary results (27), we feel that all patients who will participate in such a study should be granted the opportunity to receive infliximab, therefore a cross-over design is proposed. A cross-over design would also enhance the statistical power of the study, achieving the same statistical power with fewer patients.

Within this study, additional questions could be addressed. For example, TNF in patients with diabetes is secreted mainly by the fat cells and is involved in the development of insulin resistance and decline in the pancreatic beta-cell function. Previous studies examined the effect of anti-TNF treatment on indices of insulin resistance in non-diabetic subjects and showed that chronic treatment with anti-TNF agents may improve insulin sensitivity in humans.

The research programme will involve one country (Greece), and will include a total of 26 patients with type 1 or type 2 diabetes. The planned treatment period will be 32 weeks. Patients with clinically significant DME (i.e. BCVA < 0.4) refractory to at least two sessions of laser photocoagulation or who have leaking microaneurysms within the foveal avascular zone (FAZ) making laser photocoagulation unsafe for the central vision, will be included in the study. The study will be conducted in compliance with the protocol, ICH guidelines, Good Clinical Practice (GCP) and the applicable regulatory requirements

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to understand and sign an informed consent form.
* Signed informed consent (must be obtained before any specific procedure is performed).
* Presence of clinically significant macular edema, with visual acuity less than 0.4 corrected to EDRS scale, which is refractory to at least two sessions of laser photocoagulation, defined as: A) Thickening of the retina at or within 500 μm of the center of the macula. B) Hard exudates at or within 500 μm of the center of the macula, if associated with thickening of the adjacent retina. C) A zone or zones of retinal thickening 1 disc area or larger, any part of which is within 1 disc diameter of the center of the macula.
* Male or female aged 18-80 years, inclusive.
* Type 1 or type 2 diabetes of at least 1 year duration. Type 1 diabetes is defined clinically as a diagnosis made before the age of 36 years with a continuous need for insulin within a year of diagnosis. Type 2 diabetes is defined clinically as a diagnosis made at age of 36 or above without a need for continuous insulin therapy within a year of diagnosis.
* Postmenopausal women (no menstrual cycle for a period of a minimum of 1 year) or surgically sterilized and have a negative serum pregnancy test on entry in the study. Men must agree to use adequate birth control during the study for 6 months after the infusion of the study agent.
* Men and women of childbearing potential must use adequate birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.
* Stable diabetic therapy within the last 6 months, i.e. absence of major change in glycemic control (e.g. 2% change in HbA1c) or change in daily number of insulin injections.
* HbA1c 6.2-10%.
* The screening laboratory test must meet the following criteria: white blood cell count >5x10/L; absolute neutrophil count >1x10/L; platelet count >50x10/L; haemoglobin >100 g/L; serum creatinine <2 mg/dl; aspartate aminotransferase < 3 times the upper normal limit; alanine aminotransferase <3 times the upper normal limit; alkaline phosphatase < 2 times the upper normal limit, γ-GT< 2 times the upper normal limit
* Patients are considered eligible according to the following tuberculosis (TB) screening criteria: A)Have no history of latent or active TB prior to screening. B)Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination. C)Have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study agent. D) Within 1 month prior to the first administration of study agent, either have a negative tuberculin skin test, as outlined in appendix B, or have a newly identified positive tuberculin skin test during screening in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study agent. E)Have a chest radiograph (both posterior-anterior and lateral views), taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current active TB or old inactive TB.

Exclusion Criteria:

* Vitreoretinal traction.
* Retinal detachment.
* Proliferative diabetic retinopathy requiring immediate panretinal photocoagulation.
* Any previous eye surgery in the last 6 months before the beginning of the study (intravitreal injections are not considered ocular surgery).
* Macular Edema of ischaemic type.
* Macular Edema caused by retinal conditions other than diabetes.
* Cataract or media opacities of a degree which precludes accurate retinal photographs or OCT measurement.
* Hard exudates under the fovea.
* Uncontrolled hypertension (blood pressure above 180/110 mmHg).
* Angle closure glaucoma which precludes pharmacological dilatation of the pupil.
* Use in the previous 6 months of oral corticosteroids or in the previous month of anti-inflammatory medication.
* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last infusion) (this includes fathers who plan on fathering a child within 6 months after their last infusion).
* Have had any previous treatment with monoclonal antibodies or antibody fragments.
* History of receiving human/murine recombinant products or a known allergy to murine products. A known allergy to murine product is definitely an exclusion criterion.
* Documentation of seropositivity for human immunodeficiency virus (HIV).
* A positive test for hepatitis B surface antigen or hepatitis C virus (HCV).
* Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of the results.
* Have a known history of serious infections (e.g. hepatitis, pneumonia, or pyelonephritis) in the previous 3 months.
* Have or have had an opportunistic infection (e.g. herpes zoster, cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than tuberculosis) within 6 months prior to screening.
* Positive PPD test.
* Have a chest radiograph at screening that shows evidence of malignancy, infection, or any abnormalities suggestive of TB.
* Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (e.g. nodes in the posterior triangle of the neck, infraclavicular, epitrocheal, or periaortic area), or splenomegaly.
* Currently have a known malignancy or have a malignancy within the previous 5 years, with the exception of basal or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence.
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological or cerebral disease.
* Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access.
* Use of any investigational drug within 6 months prior to screening.
* Presence of transplanted solid organ (with the exception of corneal transplant > 3 months prior to screening).
* Have a concomitant diagnosis or history of congestive heart failure.
* Blood donation for the duration of the study
* Have allergy or other contraindication to fluorescein

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
improvement in best corrected visual acuity | 32 weeks

SECONDARY OUTCOMES:
anatomical improvement of diabetic macular edema and improvement in diabetic retinopathy | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Petros Sfikakis, MD, Principal Investigator — University of Athens
Locations (2):
- Greece (2):
  - Medical School, University of Athens, Athens
  - University of Athens, Athens

REFERENCES:
- [Derived] Sfikakis PP, Grigoropoulos V, Emfietzoglou I, Theodossiadis G, Tentolouris N, Delicha E, Katsiari C, Alexiadou K, Hatziagelaki E, Theodossiadis PG. Infliximab for diabetic macular edema refractory to laser photocoagulation: a randomized, double-blind, placebo-controlled, crossover, 32-week study. Diabetes Care. 2010 Jul;33(7):1523-8. doi: 10.2337/dc09-2372. Epub 2010 Apr 22. PMID 20413522